CLINICAL TRIAL: NCT06471933
Title: A Prospective, Single-Arm, Interventional, Multicenter, Post-Market Clinical Follow-up (PMCF) Investigation to Evaluate the Performance and Safety of Injectable Poly-LLactic Acid Dermal Filler for the Treatment of Nasolabial Fold Wrinkles
Brief Title: Post Market Clinical Follow up Evaluating the Performance and Safety of Juläine(TM) on Nasolabial Fold Wrinkles
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordberg Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOR-001
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Nasolabial Fold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Juläine (Experimental)
  Interventions: Device: Juläine

INTERVENTIONS:
Device: Juläine — Dermal filler (PLLA)

SUMMARY:
The goal of this post marketing study is to verify clincal performance and safety of CE-marked device Juläine.

The main objective is to evaluate device performance when used as intended for augmentation of shallow to deep nasolabial folds.

Participants will:

Receive 3 rounds of treatment and will be followed up for a total of 2 years.

DETAILED DESCRIPTION:
The goal of this post marketing study is to verify clincal performance and safety of CE-marked device Juläine.

The main objective is to evaluate device performance when used as intended for augmentation of shallow to deep nasolabial folds.

Participants will:

Receive 3 rounds of treatment and will be followed up for a total of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male or female, ≥18 years old.
* Immune-competent individuals.
* Presenting NLF contour deficiencies with a WSRS score between 2 (shallow wrinkle) and 4 (deep wrinkle) on both the left and right side of the face.

Exclusion Criteria:

* Having received a prior facial surgery for NLF correction, and/or received any local therapeutic treatment (e.g., dermal fillers).
* Having received in the past 2 weeks any local therapeutic treatment of the face below zygomatic arch.
* Pigmentation in NLF or having a history of hypo melanosis.
* Susceptibility to keloid formation or hypertrophic scarring.
* History of a known allergic reaction (e.g., any subject allergic to lidocaine or amide anesthetics, has a history of allergy to Gram-positive bacterial protein, or known to be allergic to any of the constituents of the product: PLLA, sodium carboxymethyl cellulose, mannitol, or sodium hyaluronate).
* History of herpes eruption, or a history of malignant skin disorder, or a history of any other serious disease.
* Hemorrhagic disease or receiving anti-coagulant therapy.
* Presenting with acute inflammation, infection, or having a history of chronic or recurrent infection potentially affecting the safety or performance of the device or increasing risk for adverse events.
* Having received in the past 2 months immunosuppressant or systemic steroid therapy.
* Having any disease that may affect wound healing, such as connective tissue disorder or serious malnutrition.
* Female who is pregnant and/or lactating
* Any other condition that as judged by the investigator may make follow-up or Investigation procedures inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Improvement on Wrinkle Severity Rating Scale (WSRS) of at least 1 grade. | 12 months after final injection
  Average improvement of at least 1 grade on the WSRS of the combined left and right NLF score.
  Score 1-5, Higher scores are a worse outcome.

SECONDARY OUTCOMES:
Percentage of subjects with improvement of at least 1 grade on the WSRS. | Up to 24 months after final injection
  Percentage of subjects with an improvement of at least 1 grade on the WSRS of the left and right (mean of the two) NLF at 3, 6 and 24 months after final injection compared to baseline (investigator assessment at all visits, blinded assessment at 12 months).
Change in WSRS score | Up to 24 months after final injection
  Change in WSRS score of the NLF at 3, 6, 12 and 24 months after final injection compared to baseline.
  Score 1-5, Higher scores are a worse outcome.
Mean WSRS of <2 at each follow-up time | Up to 24 months after final injection
  Proportion of subjects with a mean WSRS of <2 at each follow-up time point at 3, 6, 12, and 24 months after final injection.
Time to at least one grade improvement in mean WSRS and time to mean WSRS <2. | Up to 24 months after final injection
  Time to at least one grade improvement in mean WSRS and time to mean WSRS <2.
Change Face-Q score of Nasolabial Fold | Up to 24 months after final injection
  Change in FACE-Q score of the NLF at 6, 12, and 24 months after final injection compared to baseline.
  Scores 1-4: high scores better outcome
Change in Global Aesthetic in Improvement Scale | Up to 24 months after final injection
  Change in Global Aesthetic Improvement Scale (GAIS) scores evaluated by the subject, the investigator and a blinded assessor from 2D facial digital imaging at 6, 12, and 24 months after final injection compared to baseline.
  Scale 1-5; High scores worse outcome
Subject Satisfaction Scores | Up to 24 months after final injection
  Assessment of Subject Satisfaction Scores at 6, 12, and 24 months after final injection.
  Scale 1-5; High scores better outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Ribé clinic, Barcelona, Spain
- The Faculty, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to the proprietary nature of the product under investigation, which is already commercialized. Sharing participant-level data could compromise competitive advantage and intellectual property, and therefore is not aligned with the sponsor's strategic interests.